CLINICAL TRIAL: NCT04741828
Title: Persistence and Long-Term Protection of Vi Antibodies Induced by Vi-DT Conjugate Vaccines in Indonesian Adults, Adolescent, Children and Infants
Brief Title: Persistence and Long-Term Protection of Vi Antibodies Induced by Vi-DT Conjugate Vaccines in Indonesian
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: PT Bio Farma (Industry)
Collaborators: Indonesia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Typhoid 0220
Record Dates: First submitted 2021-01-27; First posted 2021-02-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Vaccine
Keywords: Vi-DT Typhoid Conjugate Vaccine

STUDY DESIGN:
Intervention Model Description: One dose Vi-DT vaccine in clinical trial subjects which is received primary dose at 6-23 months old.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vi-DT Typhoid Conjugate Vaccine (Experimental): Participants receive 1 dose (0.5ml) Vi-DT Typhoid Conjugate Vaccine, intramuscularly.
  Interventions: Drug: Vi-DT Typhoid Conjugate Vaccine

INTERVENTIONS:
Drug: Vi-DT Typhoid Conjugate Vaccine — Typhoid Conjugate Vaccine

SUMMARY:
Vi-DT Typhoid vaccine is a novel vaccine. This study will be done to know the long-term protection and persistent antibody by measured the antibody titer after 2,3,4 and 5 years after immunization.

DETAILED DESCRIPTION:
This study will be done to know the long-term protection and persistent antibody, by measured the antibody titer after 2,3,4 and 5 years after immunization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy.
* Subject who completed the phase II Vi-DT study (Typhoid 0218)
* Subjects/Parents have been informed properly regarding the study and signed the informed consent form.
* Subject/parents/legal guardians will commit to comply with the instructions of the investigator and the schedule of the trial.

Exclusion Criteria:

* Subject concomitantly enrolled or scheduled to be enrolled in another trial.
* Evolving mild, moderate or severe illness, especially infectious diseases or fever (axillary temperature ≥ 37.5oC).
* Known history of allergy to any component of the vaccines.
* History of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection.
* Any abnormality or chronic disease which according to the investigator might be compromised by the vaccination and/or interfere with the assessment of the trial objectives.

Ages: 6 Months to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 188 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
To evaluate antibody persistence 2 years after vaccination with one dose of Vi-DT in adults, adolescent, children and infants | 2 years + 2 months after primary dose
  Percentage of adults, adolescent, children and infants with seroconversion defined as >= 4 fold in antibody titer of anti Vi IgG 2 years after vaccination compared to baseline.

SECONDARY OUTCOMES:
To evaluate immunogenicity one month after booster dose of Vi-DT in subject aged 6-23 months when receiving the primary dose. | 28 days (-4/+14D)
  Percentage of subject aged 6-23 months old at primary dose with seroconversion defined as >= 4 fold in antibody titer 28 days after booster dose compared to pre booster dose.
To assess the safety following booster vaccination in subject aged 6-23 months when receiving the primary dose. | 28 days (-4/+14D)
  Percentage of subject with at least one adverse event, solicited or unsolicited, within 30 minutes, 72hours, 7 days and 28 days after booster dose.
To evaluate antibody persistence 3, 4 and 5 years after vaccination with one dose of Vi-DT in adults, adolescents, and children groups. | 5 years
  Percentage of adults, adolescents and children with seroconversion defined as ≥ 4-fold in antibody titer of anti-Vi IgG 3,4 and 5 years after vaccination compared to baseline.
To evaluate antibody persistence 1, 2 and 3 years after booster vaccination in subject aged 6-23 months when receiving the primary dose. | 3 years
  Percentage of adults, adolescents and children with seroconversion defined as ≥ 4-fold in antibody titer of anti-Vi IgG 3,4 and 5 years after vaccination compared to before booster.

CONTACTS AND LOCATIONS:
Overall Officials: Bernie E Medise, MD, Principal Investigator — Department of Child Health, School of Medicine, University of Indonesia
Locations (2):
- Indonesia (2):
  - Puskesmas Jatinegara, Jakarta
  - Puskesmas Senen, Jakarta

IPD SHARING:
Plan to Share IPD: No